CLINICAL TRIAL: NCT02061982
Title: A Non Invasive Intervention Study Performed by Subjects Themselves at Home; Evaluation of Study Infrastructure by Measuring the Effect of Caffeine on Attention and Alertness
Brief Title: Do It Yourself (DIY) Coffee Study; Test Effect of Coffee on Cognition in an at Home Setting
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: TNO (Other)
Responsible Party: Principal Investigator, W.J. Pasman, Principal Investigator, TNO
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P9568
Record Dates: First submitted 2013-11-12; First posted 2014-02-13 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: At Home Setting; Coffee With or Without Caffeine
Keywords: Do It Yourself (DIY); Caffeine; Cognition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine (Experimental): Instant coffee with or without caffeine will be provided
  Interventions: Dietary Supplement: Coffee consumption
- Coffee without caffeine (Placebo Comparator): Coffee without caffeine
  Interventions: Dietary Supplement: Coffee consumption

INTERVENTIONS:
Dietary Supplement: Coffee consumption — Coffee is consumed before cognitive tests. One cup of instant coffee with 75 mg of caffeine or 0 mg caffeine and will be prepared with 150-200 mL of hot water.
  Other Names: Instant coffee

SUMMARY:
Subjects will perform experiments in an at home-setting. The effect of caffeine in coffee will be tested in subjects with computer tests on attention and alertness. Comparison of the results with published results from controlled experiments will indicate the effectiveness of home experiments.

DETAILED DESCRIPTION:
There is increasing interest in the general public in measuring health parameters at home, instead of in a medical setting. Many tests for measuring health parameters are commonly available in drug stores as well as online. When structured, this trend may also be used for performing a randomized intervention trial.

The current study is aimed to evaluate the procedure of performing a non invasive intervention study by subjects themselves performing the tests at home.

The study is designed as a randomized, placebo-controlled, double blind, crossover study.

Subjects have to consume a cup of coffee after an overnight fast. Coffee will be prepared from instant coffee containing either regular coffee or decaff coffee. Each intervention will be given twice.

Effects on alertness and attention will be established by three computerized tests provided by Quantified Mind. The tests will be performed by the subjects at t=0 (baseline, prior to coffee consumption) and t=1h, one hour after coffee consumption, in one go. Each test will be performed during 5 minutes. During the training session the participants will be instructed to get acquainted with the task.

The evaluation of the study concerns the effect of caffeine in the at home setting versus published results, as well as reproducibility of the results.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the:

   * health and lifestyle questionnaire
2. Adult age (>18y)
3. Able to perform computerized tests
4. Voluntary participation
5. Having given written informed consent
6. Willing to comply with the study procedures
7. Moderate caffeine users
8. Able to use a desk top or laptop with internet access at home
9. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data 10 Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

1. Having a history of medical or surgical events that may significantly affect the study outcome, including attention (ADHD etc), psychological or psychiatric disorders
2. Physical, mental or practical limitations in using computerized systems
3. Use of concomitant medication including medication known for its effects on mood and/or attention (anti-depressives, sleep medication, etc)
4. Alcohol consumption > 28 units/week for males and > 21 units (drinks)/week for females
5. Personnel of TNO of location Zeist or of location Soesterberg, their partner and their first and second-generation relatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Evaluate at home tests with controlled tests in experiment in metabolic ward | 1.5 hour
  Compare results of cognitive tests in an at home setting versus the results of cognitive tests in a controlled setting in a metabolic ward. Each test costs 1.5h; there will be four test days.
  This evaluation will partly depend upon the actual number of subjects completing the tests in this at home set-up.

SECONDARY OUTCOMES:
The effect of coffee with and without caffeine on alertness and attention | 1.5 hour on four test days
  The effectiveness of the at home setting will partly be evaluated by the results found with the at home data on cognitive performance (reaction time (msec) and accuracy (% correct)).

CONTACTS AND LOCATIONS:
Overall Officials: Wilrike Pasman, PhD, Principal Investigator — Principal Investigator
Locations (1):
- TNO, Zeist, Utrecht, Netherlands

REFERENCES:
- [Derived] Pasman WJ, Boessen R, Donner Y, Clabbers N, Boorsma A. Effect of Caffeine on Attention and Alertness Measured in a Home-Setting, Using Web-Based Cognition Tests. JMIR Res Protoc. 2017 Sep 7;6(9):e169. doi: 10.2196/resprot.6727. PMID 28882811